CLINICAL TRIAL: NCT05796544
Title: Telehealth vs In-person Education for Enhancing Self-care of Ostomy Patients (SELF-STOMA): Study Design of a Non-inferiority, Randomized Controlled Trial
Brief Title: Effectiveness of Remote Self-care Education for Ostomy Patients
Acronym: SELF-STOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Ercole Vellone, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N.119.22
Record Dates: First submitted 2023-03-03; First posted 2023-04-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ostomy
Keywords: randomized controlled trial; ostomy; telehealth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a total of four remote educational sessions over 2 months.
  Interventions: Behavioral: Remote self-care education
- Control group (Active Comparator): The control group will receive the standard care, consisting of in-person standard education.
  Interventions: Behavioral: In-person self-care education

INTERVENTIONS:
Behavioral: Remote self-care education — The intervention group will receive a total of four remote educational sessions over 2 months.
  Arms: Intervention Group
Behavioral: In-person self-care education — The active comparator group will receive a total of four in-person educational sessions over 2 months.
  Arms: Control group

SUMMARY:
The primary aim of this study is to evaluate whether remote education is as effective as in-person education in improving self-care behaviors of ostomy patients.

DETAILED DESCRIPTION:
After signing the informed consent form, patients with ostomy will be assigned to the intervention or active control group (1:1). The intervention group will receive a total of four remote educational sessions over 2 months. The control group will receive the standard care, consisting of in-person standard education.

ELIGIBILITY:
Inclusion Criteria:

1. having undergone a surgical operation with subsequent ostomy placement;
2. being at least 18 years old of age;
3. absence of cognitive decline,
4. absence of any
5. being able to manage the software on the smartphone
6. be willing to participate to the trial and sign the informed consent form.

Exclusion Criteria:

1. presence of a cognitive decline, assessed with a score > 4 at the Six-item Screener
2. presence of any stomal or peristomal complication
3. not being able to read and speak Italian language

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-care maintenance | 1 month after the last intervention
  Self-care maintenance will be measured with the Ostomy Self-care Index (OSCI). Scores range from 0 to 100, with higher scores indicating better self-care maintenance

SECONDARY OUTCOMES:
Self-care monitoring | 1 month after the last intervention
  Self-care monitoring will be measured with the Ostomy Self-care Index (OSCI). Scores range from 0 to 100, with higher scores indicating better self-care monitoring
Self-care management | 1 month after the last intervention
  Self-care management will be measured with the Ostomy Self-care Index (OSCI). Scores range from 0 to 100, with higher scores indicating better self-care management
Self-care self-efficacy | 1 month after the last intervention
  Self-care self-efficacy will be measured with the Ostomy Self-care Index (OSCI). Scores range from 0 to 100, with higher scores indicating better self-care self-efficacy
Stoma-specific quality of life | 1 month after the last intervention
  Stoma-specific quality of life will be measured with the Stoma Specific Quality of Life Index- Scores on this scale range from 20 to 80, with higher scores meaning higher quality of life
Depression | 1 month after the last intervention
  Depression will be measured with the Patient Health Questionnaire 9 (PHQ-9). Scores on this scale range from 0 to 27, with higher scores indicating higher depression
Adjustment to the stoma | 1 month after the last intervention
  Adjustment to the stoma will be measured with the Stoma Adjustment Inventory-23. scores on this scale range from 0 to 92, with higher scores meaning better adjustment
Stomal and peristomal complications rates | 1 month after the last intervention
  Stomal and peristomal complications rates will be collected with a questionnaire developed by the research team.
Health care service utilization | 1 month after the last intervention
  Health care service utilization will be collected with a questionnaire developed by the research team.
Mobility (distance in km from the patient house to the hospital and vice versa, means of transportation used, and presence of a companion) | 1 month after the last intervention
  Mobility will be collected with a questionnaire developed by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Vellone, Professor, Principal Investigator — Department of Biomedicine and Prevention
Locations (5):
- Italy (5):
  - Ambulatorio infermieristico per pazienti stomizzati ASL Roma2 S.Eugenio Pertini, Roma, Rome
  - Azienda SS. Antonio e Biagio e Cesare Arrigo -, Alessandria
  - Istituto Tumori Pascale Napoli, Napoli
  - Arcispedale S. Maria Nuova Azienda ospedaliera di Reggio Emilia, Reggio Emilia
  - Tor Vergata Hospital, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] 2. Villa, G., Vellone, E., Sciara, S., Stievano, A., Proietti, M. G., Manara, D. F., ... & Pantaleo, G. (2019). Two new tools for self-care in ostomy patients and their informal caregivers: Psychosocial, clinical, and operative aspects. International Journal of Urological Nursing, 13(1), 23-30.
- [Background] Costa, A., Maria, M., Campos, C., & Santos, J. D. (2020). Effect of educational intervention in postoperative people with intestinal elimination stomies: systematic review. doi:10.6018/eglobal.19.1.368501
- [Derived] Iovino P, Vellone E, Campoli A, Tufano C, Esposito MR, Guberti M, Bolgeo T, Sandroni C, Sili A, Manara DF, Alvaro R, Rasero L, Villa G. Telehealth vs in-person education for enhancing self-care of ostomy patients (Self-Stoma): Protocol for a noninferiority, randomized, open-label, controlled trial. PLoS One. 2024 Jun 26;19(6):e0303015. doi: 10.1371/journal.pone.0303015. eCollection 2024. PMID 38924038